CLINICAL TRIAL: NCT01429480
Title: Comparison Between Two Ultrasound-guided Blocks (Transversus Abdominis Plane and Ilioinguinal/Iliohypogastric Nerve Blocks) for Pain Relief After Open Inguinal Herniorrhaphy
Brief Title: Comparison of TAP (Transversus Abdominis Plane) and Ilioinguinal/Iliohypogastric Nerve Block for Analgesia of Open Inguinal Herniorrhaphy
Acronym: TAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0065-11-HYMC
Record Dates: First submitted 2011-09-04; First posted 2011-09-07 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Pain
Keywords: Analgesia, postoperative
MeSH Terms: conditions — Pain; Agnosia | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TAP Block (Active Comparator)
  Interventions: Procedure: Preoperative Ultrasound Guided Posterior TAP Block
- II/IH Block (Active Comparator)
  Interventions: Procedure: Preoperative Ultrasound Guided Ilioinguinal/Iliohypogastric Block
- Control Group (Active Comparator)
  Interventions: Drug: Patient controlled analgesia

INTERVENTIONS:
Procedure: Preoperative Ultrasound Guided Ilioinguinal/Iliohypogastric Block
  Arms: II/IH Block
Procedure: Preoperative Ultrasound Guided Posterior TAP Block
  Arms: TAP Block
Drug: Patient controlled analgesia
  Arms: Control Group

SUMMARY:
TAP was recommended by PROSPECT for further investigation as an appropriate analgesic method after open herniorrhaphy. Ilioinguinal/iliohypogastric nerve block is one of the oldest methods of analgesia. The researchers wish to investigate whether the TAP block is as effective as the ilioinguinal/iliohypogastric nerve block?

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective primary unilateral open tension-free mesh inguinal hernia repair

Exclusion Criteria:

* Inability to consent to the study
* BMI more than 40
* Skin infection near injection site
* Chronic hepatic or renal failure
* Peripheral neuropathy
* Proven opioid dependency
* Coagulopathy
* Thrombocytopenia
* Dementia
* Lack of orientation
* Impossibility to understand VAS
* Patients suffering from chronic pain

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2011-08; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
postoperative pain | 2 days postoperatively
  Intensity of pain in rest and during movement at the operation day and 2 days postoperaive.

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

REFERENCES:
- [Derived] Stav A, Reytman L, Stav MY, Troitsa A, Kirshon M, Alfici R, Dudkiewicz M, Sternberg A. Transversus Abdominis Plane Versus Ilioinguinal and Iliohypogastric Nerve Blocks for Analgesia Following Open Inguinal Herniorrhaphy. Rambam Maimonides Med J. 2016 Jul 28;7(3):e0021. doi: 10.5041/RMMJ.10248. PMID 27487311
- See also: Related Info — http://www.postoppain.org